CLINICAL TRIAL: NCT06160128
Title: CSP #2038 - COVID-19 Pharmacotherapy Effectiveness in the VA Healthcare System (COPE-VA)
Brief Title: Clinical Outcomes and Pharmacotherapy Effectiveness in the VA Health Care System (COPE-VA)
Acronym: COPE-VA
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2038
Record Dates: First submitted 2023-11-24; First posted 2023-12-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: COVID-19, SARS-CoV-2 Infection; RSV; Influenza
Keywords: COVID-19; pharmacotherapy effectiveness; SARS-CoV-2; antiviral; RSV; influenza; respiratory viruses
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: None Retained — none collected or retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Outpatient Veterans with risk factors for severe COVID-19 & tested positive during Jan-Feb 2022: This cohort study assessed outpatient Veterans with risk factors for severe COVID-19 who tested positive for SARS-CoV-2 during January and February 2022.
  The purpose is to describe factors associated with receipt of outpatient COVID-19 pharmacotherapies in the Veterans Affairs (VA) health care system.
- Nonhospitalized Veterans in VHA at risk for SARS-CoV-2 Jan-Jul 2022: Three retrospective target trial emulation studies comparing matched cohorts of nirmatrelvir-ritonavir versus no treatment, molnupiravir versus no treatment, and nirmatrelvir- ritonavir versus molnupiravir.
  The purpose is to measure the effectiveness of nirmatrelvir-ritonavir and molnupiravir for outpatient treatment of COVID-19.
- Outpatient Veterans who tested positive for SARS-CoV-2 from Jan 2022 through Jan 2023: This cohort study evaluated nonhospitalized Veterans in VHA care who tested positive for SARS-CoV-2 from January 2022 through January 2023 using VHA and linked Community Care and Medicare databases.
  The purpose is to analyze trends and factors associated with prescription of outpatient COVID-19 pharmacotherapies within the Veterans Health Administration (VHA).
- Outpatient Veterans with risk factors for severe COVID-19 & tested positive during Jan-Jul 2022: Retrospective target trial emulation study comparing matched cohorts receiving nirmatrelvir-ritonavir versus no treatment.
  The purpose is to measure the effectiveness of outpatient treatment of COVID-19 with nirmatrelvir-ritonavir in preventing Post COVID conditions.

SUMMARY:
The purpose of this study is to comprehensively describe the temporal and geographic utilization of COVID-19 therapies used for mild to moderate disease during different periods of SARS-CoV-2 variant circulation as well as to compare demographic and clinical characteristics of Veterans who are treated or do not receive these different therapies. The investigators will also perform similar descriptive epidemiology for other respiratory viruses, including RSV and influenza and other infectious diseases. This first phase will critically inform feasibility and direction of the second phase, in which the investigators will use target trial emulation design to study the comparative effectiveness of therapies and vaccines for COVID-19, respiratory viruses, including RSV, and influenza, and other infectious diseases.

DETAILED DESCRIPTION:
Objectives:

This study will be completed in two phases. In the first phase, the investigators will establish a source population and comprehensively describe the temporal and geographic utilization of COVID-19 pharmacotherapies beginning July 2021. These therapies include casirivimab and imdevimab, bamlanivimab and etesevimab, sotrovimab, nirmatrelvir, molnupiravir, and remdesivir. The investigators will also compare demographic and clinical characteristics of Veterans who are treated or do not receive these therapies. Phase 1 will inform the study design and analytic protocol of Phase 2. Phase 1 will also inform critical policy questions and national guidance regarding COVID-19 pharmacotherapies in the VA healthcare system with the potential to inform policy across other healthcare systems.

In the second phase, the investigators will conduct target trial emulation studies to determine the effectiveness and comparative effectiveness of current pharmacotherapies for COVID-19 in preventing short- and long-term adverse outcomes related to SARS-CoV-2 infection. The investigators will use a sequence of comparative effectiveness studies through emulation to help establish a common framework sharing a similar population, design, and outcomes for a rapid-response, adaptive observational study design to characterize utilization and determine the effectiveness and comparative effectiveness of novel therapeutic agents authorized for the treatment of mild to moderate COVID-19 in Veterans. Phase 2 will provide an infrastructure upon which subsequent observational studies can be performed, which will include other infectious diseases of interest, ultimately ensuring the timeliness and pertinence of VA research.

Research Design and Methodology:

In the first phase, the investigators will conduct a descriptive, retrospective, electronic health record-based study among Veterans aged 18 years with a laboratory-confirmed positive test for SARS-CoV-2 or a diagnosis of COVID-19 documented at any time since the beginning of the pandemic in January 2020 to present. The investigators will describe the geographic distribution (by VISN, state, and distance from place of residence to the closest VAMC and/ COVID-19 infusion facilities) of Veterans receiving each of the COVID-19 antiviral and monoclonal antibody therapies during different periods of SARS-CoV-2 variant circulation (i.e., January 1, 2022, to present for Omicron). The investigators will also compare baseline demographic characteristics, clinical characteristics including underlying medical conditions and prior SARS-CoV-2 infections, SARS-CoV-2 vaccination status, National Institutes of Health (NIH) risk group tiers for prioritization of treatments, concurrent outpatient medications, and time from positive test to treatment among Veterans receiving different antiviral and monoclonal antibody therapies as well as eligible Veterans who are not treated during different periods of SARS-CoV-2 variant circulation. This established framework will also be used to identify Veterans who tested positive for other respiratory viruses, including influenza virus or respiratory syncytial virus (RSV), and other infectious diseases in the same time period and describe their characteristics, risk factors and treatments.

In the second phase, the investigators will conduct retrospective and prospective target trial emulation studies to evaluate the effectiveness and comparative effectiveness of different pharmacotherapies for mild-to-moderate COVID-19 in patients with documented SARS-CoV-2 infection by period of predominant SARS-CoV-2 variant circulation. The established framework will be used to investigate vaccine and pharmacotherapy effectiveness for SARS-CoV-2 and other respiratory viruses, including influenza and respiratory syncytial virus (RSV) and other infectious diseases using observational data from the VHA electronic health records.

Impact Significance:

Data on real-world utilization and clinical outcomes in the Veteran population are needed to inform clinical, operational and research partners in the VA and other healthcare systems on strategies for optimizing the utilization of pharmacotherapies and vaccines against COVID-19 and other infectious diseases. Ongoing evaluations will be essential as new variants emerge, vaccination practices evolve, and new pharmacotherapies are introduced. This study will establish a common framework sharing a similar population, design, and outcomes for a rapid-response, adaptive platform observational study design to characterize utilization and determine the effectiveness and comparative effectiveness of novel therapeutic agents authorized for the treatment of mild to moderate COVID-19, respiratory viruses, including RSV and influenza, and other infectious diseases in Veterans.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

- Veterans aged 18 years with a laboratory-confirmed positive test for SARS-CoV-2 or a diagnosis of COVID-19 documented at any time since the beginning of the pandemic in January 2020 to present.

Phase 2:

* All Veterans aged 18 years alive and in VHA care as of January 2018.
* Specific exclusion/inclusion criteria and observation periods will be further defined for each sub-study (See outcomes/publications).

Exclusion Criteria:

* VA employees who are not enrollees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: VA enrollees infected from January 1, 2022 through February 28, 2022 as an example. Subsequent trials will be executed as the pandemic evolves
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Receipt of any COVID-19 pharmacotherapy, including sotrovimab, nirmatrelvir boosted with ritonavir, molnupiravir, or remdesivir | January and February 2022
  The odds of receipt of any COVID-19 pharmacotherapy, including sotrovimab, nirmatrelvir boosted with ritonavir, molnupiravir, or remdesivir were estimated using multivariable logistic regression
Incidence of any hospitalization or all-cause mortality at 30 days and from 31 to 180 days | January through July 2022
  Three retrospective target trial emulation studies comparing matched cohorts of nirmatrelvir-ritonavir versus no treatment, molnupiravir versus no treatment, and nirmatrelvir- ritonavir versus molnupiravir.
Monthly receipt of any COVID-19 pharmacotherapy (nirmatrelvir-ritonavir, molnupiravir, sotrovimab, or bebtelovimab) | January 2022 through January 2023
  To analyze trends and factors associated with prescription of outpatient COVID-19 pharmacotherapies within the Veterans Health Administration (VHA).
Cumulative incidence of 31 potential PCCs at 31 -180 days after treatment or a matched index date, including cardiac, pulmonary, renal, thromboembolic, gastrointestinal, neurologic, mental health, musculoskeletal, endocrine, and general conditions | January through July 2022
  Retrospective target trial emulation study comparing matched cohorts receiving nirmatrelvir-ritonavir versus no treatment.
Incidence of any hospitalization or all-cause mortality at 30 days | April 2022 through March 2023
  target trial emulation study in the Veterans Health Administration comparing nirmatrelvir-ritonavir treated versus matched untreated Veterans at risk for severe COVID-19 who tested positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
Prediction of 30-day COVID-19 hospitalization and death in the Omicron era for contemporary clinical and research applications | March 1, 2022, and March 31, 2023
  Full models incorporated 84 predictors, including demographics, comorbidities, and receipt of COVID-19 vaccinations and anti-SARS-CoV-2 treatments. Parsimonious models included 19 predictors. We created models for 30-day hospitalization or death, 30-day hospitalization, and 30-day all-cause mortality. We used the Super Learner ensemble machine learning algorithm to fit prediction models. Model performance was assessed with the area under the receiver operating characteristic curve (AUC), Brier scores, and calibration intercepts and slopes in a 20% holdout dataset.
RSVPreF3 or RSVpreF vaccination compared with no RSV vaccination for the prevention of documented RSV infection and associated health-care use among Veterans | March 1, 2022, and March 31, 2023
  The primary outcome was any positive RSV test result occurring from day 14 following the index date until the end of the study period.7,8 Secondary outcomes included RSV-associated emergency department or urgent care encounters, RSV-associated acute hospitalisations, RSV associated intensive care unit (ICU) admissions, and death. RSV-associated health-care encounters were defined as any corresponding encounter occurring the day before until 1 day after the eligible positive RSV test result. Death was defined as any death occurring on the day of until 30 days after the eligible positive RSV test result.
compare disease severity of COVID-19, influenza, and RSV among US Veterans | August 1, 2022, and March 31, 2023, or between August 1, 2023, and March 31, 2024.
  This retrospective cohort study analyzed national US Veterans Health Administration electronic health record data of nonhospitalized Veterans who underwent same-day testing for SARS-CoV-2, influenza, and RSV, and were diagnosed with a single infection between August 1, 2022, and March 31, 2023, or between August 1, 2023, and March 31, 2024.
  Following inverse probability weighting, the cumulative incidence and risk differences (RDs) were calculated for the primary outcomes of 30-day hospitalization, intensive care unit admission, and death, as well as the secondary outcome of long-term death extending through 180 days.
Determine XBB.1.5 COVID-19 VE and the extent to which it declines over time | October 2,2023- January 3, 2024
  Outcomes were ascertained through 10 May 2024 and included any positive result on a SARS-CoV-2 test from day 10 after the matched index date, subsequent hospitalization within 1 day before or 10 days after the positive result, or death within 30 days after the positive result. Vaccine effectiveness was estimated as 100x (1-risk ratio).
Determine if severe SARS-CoV-2 infection increases risk of selected PCCs or death up to 1 year after infection in wild-type (WT), Alpha-transition, Delta, and Omicron eras | March 2020 and April 2022
  Investigated whether severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection increases the risk of selected PCCs or death up to 1 year after infection, separately in the wild-type (WT), Alpha-transition, Delta, and Omicron eras and by vaccination status.
Determined budget cost of providing nirmatrelvir-ritonavir to Veterans with COVID-19 on 30-day healthcare costs to inform procurement strategies in large healthcare systems | April 2022 through March 2023
  The decision tree analysis included transition states from cohort entry (ie, infection and treatment) to ED visit, hospitalization without ICU admission, hospitalization with ICU admission, recovery, and death (Figure 1). Decision trees were created for each subgroup and treatment allocation and parameterized with subgroup and treatment specific transition probabilities. In total, 26 trees (13 subgroups and 2 treatment scenarios) were created and parameterized with over 150 transition probabilities.
Evaluate the impact of different time zero designations on results and inferences from a cohort study comparing the effectiveness of nirmatrelvir ritonavir treatment versus no COVID-19 antiviral treatment in preventing 30-day hospitalization and death | April 2022-March 2023
  Identified US Veterans who tested positive for SARS-CoV-2 from April 2022-March 2023 and compared nirmatrelvir-ritonavir versus no treatment using 5 time zero approaches: test-date (treated) versus test-date (untreated) with matching allowing treatment on days 0-5 (approach 1a) or day 0 only (1b), test-date versus test-date with a clone-censor-weight method (1c), treatment date versus test-date (2) with matching, or treatment date versus matched index date (3).
Asses the long-term effectiveness of a single respiratory syncytial virus (RSV) vaccine dose against RSV illness and associated health care use | September 2023 to March 2024.
  The primary outcome was any positive RSV test result from day 14 following the matched index date. Secondary outcomes included RSV-associated emergency department or urgent care visits, hospitalizations, or intensive care unit admissions. Vaccine effectiveness was estimated as 100 × (1 - risk ratio).
Estimate the long-term vaccine effectiveness (VE) of the 2024-2025 COVID-19 vaccines targeting the KP.2 Omicron variant within the Veterans Health Administration | August 1, 2024- April 12, 2025
  Vaccine effectiveness against documented SARS CoV-2 infection, SARS-CoV-2 associated ED/UC visit, SARS-CoV-2 associated hospitalization or SARS-CoV-2 associated death

CONTACTS AND LOCATIONS:
Overall Officials: Kristina L Bajema, MD, Study Chair — VA Portland Health Care System, Portland, OR; George N. Ioannou, MD MS, Study Chair — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available